CLINICAL TRIAL: NCT03547492
Title: Developmental Intervention for Infants of Adolescent Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB Net ID 792482-3
Record Dates: First submitted 2018-05-24; First posted 2018-06-06 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Development, Child; Adolescent Behavior; Language Development; Language Delay
Keywords: language; LENA; adolescent
MeSH Terms: conditions — Adolescent Behavior; Language Development Disorders; Language

STUDY DESIGN:
Intervention Model Description: Random assignment to language (intervention) or motor (control) focused curriculums
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Language Intervention (Experimental): 1. Baseline LENA recording 2. Review language curriculum and motor curriculum with study personnel 2. Direct linguistic feedback of baseline LENA recording 4. 2nd LENA recording completed and analyzed 5. Direct or mailed linguistic feedback of 2nd LENA recording 6. 16- Weekly text messages 7. 4 month LENA recording with mailed linguistic feedback 8. 12 month LENA recording with mailed linguistic feedback
  Assessments:
  1. Ages and Stages Questionnaire at 4 and 12 months
  2. Maternal Peabody Picture Vocabulary test at 4 months
  3. Edinburgh Post-partum Depression Scale at 4 months
  4. MacArthur Bates Communicative Developmental Inventory: Words and Gestures at 12
  Participants receive a book at each interaction.
  Interventions: Behavioral: Teaching Talking; Behavioral: LENA recordings-language; Behavioral: Mastering Movement; Behavioral: Language text messages; Behavioral: Motor text messages
- Motor Control (Active Comparator): 1. Baseline LENA recording
  2. Review motor curriculum with study personnel
  3. 2nd LENA recording completed and analyzed
  4. 4- monthly text messages
  5. 4 month LENA recording
  6. 12 month LENA recording with mailed linguistic feedback of all recordings
  Assessments:
  1. Ages and Stages Questionnaire at 4 and 12 months
  2. Maternal Peabody Picture Vocabulary test at 4 months
  3. Edinburgh Post-partum Depression Scale at 4 months
  4. MacArthur Bates Communicative Developmental Inventory: Words and Gestures at 12
  Participants receive a toy at each interaction.
  Interventions: Behavioral: LENA recordings-motor; Behavioral: Mastering Movement; Behavioral: Motor text messages

INTERVENTIONS:
Behavioral: Teaching Talking — Written packet including 8 lessons: What's My Corrected Age, Watch Me Learn (language milestones in the 1st year of life), Reading Aloud, Sing-a-long: Sleepy Songs, Sing-a-long: Alert Songs, Copying First Sounds, Playing Games, Talk to Your Baby.
  Arms: Language Intervention
Behavioral: LENA recordings-language — LENA a special recording device. It records for 16 hours inside a specially designed infant vest. The recording is analyzed by a computer that generates an output of total number of adult words, infant vocalizations and conversational turns during the recording period. 4 LENA recordings are obtained: baseline, after reviewing Teaching Talking and linguistic feedback of first recording, 4 and 12 months of age. Participants are mailed feedback of their 2nd, 4 and 12 month recordings.
  Arms: Language Intervention
Behavioral: LENA recordings-motor — LENA a special recording device. It records for 16 hours inside a specially designed infant vest. The recording is analyzed by a computer that generates an output of total number of adult words, infant vocalizations and conversational turns during the recording period. 4 LENA recordings are obtained: baseline, 2nd, 4 and 12 months of age. Participants are mailed feedback on recordings after completing study.
  Arms: Motor Control
Behavioral: Mastering Movement — A written curriculum containing 5 lessons adopted from Beautiful Beginnings: What's My Corrected Age, Watch Me Move! (review of motor milestones in 1st year), Gentle Stretching and Exercise, Tummy Time, Help Me Learn to...
Behavioral: Language text messages — 12 weekly text messages. Each is 1-2 sentences to review concepts of Teaching Talking
  Arms: Language Intervention
Behavioral: Motor text messages — 4 text messages sent every 4 weeks. Each is 1-2 sentences reviewing concepts of Mastering Movement

SUMMARY:
This is a randomized control trial to evaluate a simple language intervention curriculum that utilizes LENA recordings, linguistic feedback and text-message review of content to improve language environments and outcomes for infants with adolescent mothers.

DETAILED DESCRIPTION:
Mother-infant pairs are enrolled while in the hospital after birth. Enrolled participants are randomized into a language (intervention) or motor (control) group. All participants have a baseline LENA (device that captures 16 hour recording and associated computer analysis generates a report of numbers of adult words spoken, infant vocalization and conversational turns). Interventions after the baseline recording by group are as follows:

Intervention:

1. Review language curriculum and motor curriculum with study personnel
2. Direct linguistic feedback of baseline LENA recording
3. 2nd LENA recording completed and analyzed
4. Direct or mailed linguistic feedback of 2nd LENA recording
5. 16- Weekly text messages
6. 4 month LENA recording with mailed linguistic feedback
7. 12 month LENA recording with mailed linguistic feedback

Control:

1. Review motor curriculum with study personnel
2. 2nd LENA recording completed and analyzed
3. 4- monthly text messages
4. 4 month LENA recording
5. 12 month LENA recording with mailed linguistic feedback of all recordings

Both groups undergo the following assessments:

1. Ages and Stages Questionnaire at 4 and 12 months
2. Maternal Peabody Picture Vocabulary test at 4 months
3. Edinburgh Post-partum Depression Scale at 4 months
4. MacArthur Bates Communicative Developmental Inventory: Words and Gestures at 12

ELIGIBILITY:
Inclusion Criteria:

* Infants ≥30 weeks born to 15-20 year old mothers

Exclusion Criteria:

* Congenital anomalies associated with adverse developmental outcomes
* Non-English speaking mothers
* No cell phone
* Mother not available for follow-up
* State custody of mother or infant.

Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2013-01-25 (Actual); Primary Completion 2015-11-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
MacArthur CDI | 12 months
  MacArthur Bates Communicative Developmental Inventory: Words and Gestures scores

SECONDARY OUTCOMES:
LENA Counts | birth, 4 months, 12 months
  Adult word counts, conversational turns and infant vocalization of each LENA recording
Ages & Stages Questionnaire | 4 months, 12 months
  Parent report of development at 4 and 12 months of age

IPD SHARING:
Plan to Share IPD: No
IPD will not be made available to other researchers

REFERENCES:
- [Background] Caskey M, Stephens B, Tucker R, Vohr B. Importance of parent talk on the development of preterm infant vocalizations. Pediatrics. 2011 Nov;128(5):910-6. doi: 10.1542/peds.2011-0609. Epub 2011 Oct 17. PMID 22007020
- [Background] Squires J, Bricker D, Potter L. Revision of a parent-completed development screening tool: Ages and Stages Questionnaires. J Pediatr Psychol. 1997 Jun;22(3):313-28. doi: 10.1093/jpepsy/22.3.313. PMID 9212550
- [Background] Thal D, Desjardin JL, Eisenberg LS. Validity of the MacArthur-Bates Communicative Development Inventories for measuring language abilities in children with cochlear implants. Am J Speech Lang Pathol. 2007 Feb;16(1):54-64. doi: 10.1044/1058-0360(2007/007). PMID 17329675